CLINICAL TRIAL: NCT05295433
Title: A Phase 1/2, Global, Open-Label, Extension Study to Evaluate the Long-Term Safety and Clinical Activity of mRNA-3705 in Participants Previously Enrolled in Other Clinical Studies of mRNA-3705
Brief Title: An Extension Study to Evaluate the Long-Term Safety and Clinical Activity of mRNA-3705 in Participants Previously Enrolled in Other Clinical Studies of mRNA-3705
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-3705-P101-EXT; 2021-000446-17 (EudraCT Number); 2022-501997-20-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-02-14; First posted 2022-03-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Methylmalonic Acidemia
Keywords: Isolated Methylmalonic acidemia; Isolated methylmalonic aciduria; Elevated methylmalonic acid (MMA); Metabolism, Inborn Errors; Genetic Diseases; Moderna; mRNA; mRNA-3705
MeSH Terms: conditions — Methylmalonic acidemia; Metabolism, Inborn Errors; Genetic Diseases, Inborn | interventions — Methylmalonyl-CoA Mutase

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- mRNA-3705 (Experimental): Participants will receive mRNA-3705 at the same dose levels at the same dosing interval (every 2 weeks [Q2W], or every 3 weeks [Q3W]) last received in the clinical study of mRNA-3705 in which they initially participated, unless the Sponsor recommends modification.
  Interventions: Drug: mRNA-3705

INTERVENTIONS:
Drug: mRNA-3705 — A sterile liquid for injection
  Other Names: modified mRNA encoding human; methylmalonyl-coenzyme A mutase

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and clinical activity of mRNA-3705 administered to participants with isolated methylmalonic acidemia (MMA) due to methylmalonyl-coenzyme A mutase (MUT) deficiency who have previously participated in other clinical studies of mRNA-3705.

DETAILED DESCRIPTION:
Participants with isolated MMA due to MUT deficiency who were previously enrolled in other clinical studies of mRNA-3705 will have the option to enroll into this extension study provided all eligibility criteria have been met. The study will include 2 periods: 1) Treatment Period and 2) Follow-up Period (up to 6 months after the last dose of study drug).

Treatment Period will continue unless one of the following occurs: mRNA-3705 receives marketing approval and reimbursement in the country of origin of the participant (following market approval and access being in place, all participants who wish to continue treatment will be offered mRNA-3705 through market access, with the intention of preventing treatment interruption. Other appropriate access program is offered as allowed by local regulation to continue treatment with mRNA-3705. Safety monitoring will be performed for all participants under treatment per market access requirements), the participant discontinues study drug, the participant is no longer receiving clinical benefit in the opinion of the Investigator, or Sponsor discontinues the development of mRNA-3705.

ELIGIBILITY:
Inclusion Criteria:

* Completed the assigned dose regimen treatment time period in other clinical studies of mRNA-3705 or is eligible for early transition to this study because they missed more than 3 consecutive doses of study drug due to coronavirus disease 2019 (COVID-19) vaccination during Study mRNA-3705-P101 Part 1.
* Completed the End of treatment (EOT) Visit (or End of Study Visit in the case of unscheduled dosing) in Study mRNA-3705-P101 within 10 days of their first dose of mRNA-3705 in this extension study.

Exclusion Criteria:

* Not expected to receive clinical benefit from continued mRNA-3705 administration, in the opinion of the Investigator.
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the Investigator, may put the individual at increased risk by participating in this study.
* History of liver and/or kidney transplant.

NOTE: Other inclusion and exclusion criteria may apply.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2034-04-02 (Estimated); Study Completion 2034-04-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Drug-Related TEAEs, Unrelated TEAEs, Adverse Events of Special Interests (AESIs), Serious Adverse Events (SAEs) and TEAEs Leading to Discontinuation | Baseline up to follow-up period (up to 6 years + 6 months)

SECONDARY OUTCOMES:
Percent Change in Plasma Methylmalonic Acid and 2-Methylcitric Acid (2-MC) Levels (Primary Biomarkers) From Baseline up to 18 Months | Baseline, Year 6 (Treatment Period) + Month 6 (Follow up)
Pre- and Postdose Human Methylmalonyl-Coenzyme A Mutase (hMUT) mRNA and SM-86 Levels | Baseline up to 6 years
Change From Baseline in Pretreatment and Post-treatment Annualized Metabolic Decompensation Events (MDEs) Rate | Baseline, Year 6 (Treatment Period) + Month 6 (Follow up)
Number of Healthcare Resource Utilization Visits | Baseline up to Year 6 (Treatment Period) + Month 6 (Follow up)
Number of Annualized MMA-related Hospitalizations | Baseline up to Year 6 (Treatment Period) + Month 6 (Follow up)
Number of Annualized MMA-related Healthcare Visits | Baseline up to Year 6 (Treatment Period) + Month 6 (Follow up)
Number of Anti-Polyethylene Glycol (PEG) and Anti-hMUT Antibodies | Baseline up to Year 6 (Treatment Period) + Month 6 (Follow up)
Change in Health-Related Quality of Life (HRQoL) as Measured Using the Pediatric Quality of Life Inventory (PedsQL™) at Month 3 up to 18 Months | Month 3, Year 6 (Treatment Period) + Month 6 (Follow up)
Change in Investigator Global Assessment of Improvement (IGA-I) Score | Baseline up to Year 6 (Treatment Period) + Month 6 (Follow up)
Change in Investigator Global Assessment of Severity (IGA-S) Score | Baseline up to Year 6 (Treatment Period) + Month 6 (Follow up)
Change in EuroQoL 5-Dimensions 5-level/Youth Questionnaire (EQ-5D-5L/Y) Score | Baseline up to Year 6 (Treatment Period) + Month 6 (Follow up)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Altman Clinical and Translational Research Institution, San Diego, California
- Canada (2):
  - Stollery Children's Hospital University of Alberta, Edmonton, Alberta
  - Hospital For Sick Children, Toronto, Ontario
- Hôpital Necker - Enfants Malades APHP, Paris, France
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (2):
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Royal Manchester Childrens Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Undecided